CLINICAL TRIAL: NCT03519568
Title: Evaluating Immunogenicity and Safety Effect on Combined Immune Effect of EV71 Inactivated Vaccine and HepB、MPSV-A、MR、JE-L：A Multi-center Randomized Controlled Trial
Brief Title: Clinical Study on Combined Immune Effect of EV71 Inactivated Vaccine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Province Centers for Disease Control and Prevention (Other)
Collaborators: Hunan Provincial Center for Disease Control and Prevention (Other); Shaanxi Provincial Center for Disease Control and Prevention (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ShandongCDCP
Record Dates: First submitted 2018-03-25; First posted 2018-05-09 (Actual); Last update posted 2018-05-09 (Actual); Status verified 2018-04

CONDITIONS: Enterovirus 71 Inactivated Vaccine; HFMD

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Combination inoculation group (Experimental): GroupⅠ: HepB:3 and EV71 were injected at 6 months old, EV71 second dose was injected at 7 months old GroupⅡ: MPSV-A:1 and EV71 were injected at 6 months old, EV71 second dose was injected at 7 months old, MPSV-A:1 second dose was injected at 9 months old GroupⅢ: MR and EV71 were injected at 8 months old, EV71 second dose was injected at 9 months old GroupⅣ: JE-Land EV71 were injected at 8 months old, EV71 second dose was injected at 9 months old
  Interventions: Biological: EV71 (inoculation vaccine)
- Separate inoculation control group (Active Comparator): GroupⅠ: HepB:3 third dose was injected at 6 months old GroupⅡ: MPSV-A:1 was injected at 6 months old, then MPSV-A:1 second dose was injected at 9 months old GroupⅢ: MR was injected at 8 months old GroupⅣ: JE-L was injected at 8 months old
  Interventions: Biological: EV71 (inoculation vaccine)
- EV71 inoculation control group (Active Comparator): GroupⅠ: EV71 was injected at 8 months old, then EV71 second dose was injected at 9 months old GroupⅡ: EV71 was injected at 8 months old, then EV71 second dose was injected at 9 months old GroupⅢ: EV71 was injected at 8 months old, then EV71 second dose was injected at 9 months old GroupⅣ: EV71 was injected at 8 months old, then EV71 second dose was injected at 9 months old
  Interventions: Biological: EV71 (inoculation vaccine)

INTERVENTIONS:
Biological: EV71 (inoculation vaccine) — EV71 vaccine 0.5ml per dose, Wuhan Biological Products Co., Ltd., Wuhan, Hubei Province, China 10μg HepB 0.5ml per dose, Wuhan Biological Products Co., Ltd., Wuhan, Hubei Province, China 30ug MPSV-A 0.5ml per dose, Wuhan Biological Products Co., Ltd., Wuhan, Hubei Province, China MR 0.5ml per dose, Beijiing Biological Products Co., Ltd., Beijing, China JE-L 0.5ml per dose, Chengdu Biological Products Co., Ltd., Chengdu,Sichuan Province, China

SUMMARY:
Background: To prevent and control the epidemic of HFMD and related diseases caused by EV71 infection, the development of EV71 vaccine has been developed in many countries or regions. According to the requirements of drug registration approval, we need to evaluate immunogenicity and safety effect on combined immune effect of EV71 inactivated vaccine and other vaccines (HepB、MPSV-A、MR、JE-L).

Method: Four experimental groups (HepB:3+EV71, MPSV-A:1+EV71, MR+EV71, JE-L+EV71) were included in this clinical trail. In addition to the meningococcal vaccine research group, the other three groups were followed up for the 4 times. The initial blood samples were collected, and the first dose vaccine was inoculated at the same time. EV71 second doses of vaccine were inoculated at 30 day, the blood was collected after 30 days of immunization with second doses. 6 months of safety follow-up was carried out in the whole clinical trial after vaccination. The meningococcal vaccine research group increased 1 follow-up after the second dose of MPSV-A vaccine. The index of immunogenicity and safety effect in four experimental groups need to be evaluated.

DETAILED DESCRIPTION:
Study design and participants The study was conducted in four provinces (Shandong, Shanxi, Shaanxi and Hunan) of China, which contains Haiyang city, Rushan city, Shimen County, Chen Cang District, Qishan County, Taigu County and Qi County. 6/8 months children were recruited in this study, individuals were randomly assigned to experimental group and control group. Demographic information (age, sex, height and weight) was made and blood samples were collected for each individual in the same way.

Vaccine inoculation and follow-up

TestⅠ(HepB:3+EV71):

Experimental group - 6 month old HepB third dose and EV71 first dose were inoculated at the same time, 7 month old EV71 second dose was inoculated, blood samples from the participants were collected at 8 month old; Control group 1- 6 month old HepB third dose was inoculated separately, blood samples from the participants were collected after two months; Control group 2 - 6 month old EV71 first doses was inoculated, 7 month old EV71 second dose was inoculated, blood samples from the participants were collected at 8 month old.

TestⅡ(MPSV-A:1+EV71):

Experimental group - 6 month old MPSV-A first dose and EV71 first dose were inoculated at the same time, 7 month old EV71 second dose was inoculated, 9 month old MPSV-A second dose was inoculated, blood samples from the participants were collected at 10 month old; Control group 1- 6 month old MPSV-A first dose was inoculated separately, 9 month old MPSV-A second dose was inoculated separately, blood samples from the participants were collected at 10 month old; Control group 2 - 6 month old EV71 first doses was inoculated, 7 month old EV71 second dose was inoculated, blood samples from the participants were collected at 10 month old.

TestⅢ (MR+EV71):

Experimental group - 8 month old MR first dose and EV71 first dose were inoculated at the same time, 9 month old EV71 second dose was inoculated, blood samples from the participants were collected at 10 month old.

Control group 1- 8 month old MR first dose was inoculated separately, blood samples from the participants were collected at 10 month old; Control group 2 - 8 month old EV71 first doses was inoculated, 9 month old EV71 second dose was inoculated, blood samples from the participants were collected at 10 month old.

TestⅣ(JE-L+EV71):

Experimental group - 8 month old JE-L first dose and EV71 first dose were inoculated at the same time, 9 month old EV71 second dose was inoculated, blood samples from the participants were collected at 10 month old.

Control group 1- 8month old JE-L first dose was inoculated separately, blood samples from the participants were collected at 10 month old; Control group 2 - 8 month old EV71 first doses was inoculated, 9 month old EV71 second dose was inoculated, blood samples from the participants were collected at 10 month old.

EV71 vaccine 0.5ml per dose, Wuhan Biological Products Co., Ltd., Wuhan, Hubei Province, China; 10μg HepB 0.5ml per dose, Wuhan Biological Products Co., Ltd., Wuhan, Hubei Province, China; 30ug MPSV-A 0.5ml per dose, Wuhan Biological Products Co., Ltd., Wuhan, Hubei Province, China; MR 0.5ml per dose, Beijiing Biological Products Co., Ltd., Beijing, China; JE-L 0.5ml per dose, Chengdu Biological Products Co., Ltd., Chengdu,Sichuan Province, China Immunogenicity end point Detection of serum antibody EV71 vaccine by culture neutralization test, the definition of positive for neutralizing antibody titers of <1:8 before inoculation, inoculation after neutralizing antibody titers than 1:8; or before inoculation neutralizing antibody titer is above 1:8, the titer of neutralizing antibody after vaccination appeared more than 4 times the growth.

Hepatitis B vaccine seroconversion was defined as Anti-HBs<10mIU/ml before inoculation, Anti-HBs after inoculation was more than 10mIU/ml.

Leprosy vaccine using measles rubella immunoglobulin ELISA detection test, measles >200U/ml positive for rubella >20U/ml positive or positive before inoculation; after inoculation, antibody positive growth is more than 4 times.

Japanese encephalitis vaccine serum samples by using PRNT test before immunization antibody titer after inoculation was less than 1:5, at 1:10, or after vaccination antibody titer than before inoculation is no less than 4 times of growth is positive.

Meningococcal vaccine samples A meningococcal bactericidal antibody level in serum by micro bactericidal antibody test, the antibody titer after inoculation than before inoculation is no less than 4 times of growth is positive.

Safety assessment Safety assessment Participants were provided with diary cards to record the occurrence and severity of solicited local reactions at the injection site (pain, induration, erythema, edema, pruritus) during 7 days after vaccination, solicited systemic reactions (fever, headache, fatigued, cough, myalgia, asthenia, vertigo, diarrhea), and any unsolicited adverse during 29 days after vaccination.

Statistical analyses The quantitative index lists the standard deviation, the median, the maximum and the minimum, and the qualitative index or the grade index list the frequency distribution table. The antibody titers of immunogenicity index should be represented by geometric mean, median, maximum and minimum value and 95% confidence interval. The antibody titer should be analyzed by logarithmic transformation.

A list of the total population, susceptible and non susceptible seroconversion rate and 95% confidence interval, and calculation (test group and control group) rate difference and 95% confidence interval, non-inferiority test; the test group and the control group between the antibody geometric mean (GMT/GMC) compared with the t test after logarithmic transformation P, with less than 0.05 as there were statistically significant differences in the standard

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for group Ⅰ（HepB:3+EV71）were as follows:

1. aged ≥ 6 months
2. sign the informed consent form
3. the legal guardians participate in all the planned follow-up and be able to comply with all research procedures
4. the subjects have completed the basic immunization of 2 needle recombinant hepatitis B vaccine, there is no inoculation history of EV71 vaccine, and no history of EV71 infection
5. the last vaccination intervals ≥ 14 days
6. temperature ≤ 37℃

Inclusion criteria for group Ⅱ（MPSV-A:1+EV71）were as follows:

1. aged ≥ 6 months
2. sign the informed consent form
3. the legal guardians participate in all the planned follow-up and be able to comply with all research procedures
4. there is no inoculation history of EV71 vaccine, and there is no history of EV71 infection
5. the last vaccination intervals ≥ 14 days
6. temperature ≤ 37℃

Inclusion criteria for group Ⅲ（MR+EV71）were as follows:

1. aged ≥ 8 months
2. sign the informed consent form
3. the legal guardians participate in all the planned follow-up and be able to comply with all research procedures
4. there is no inoculation history of EV71 vaccine, and there is no history of EV71 infection
5. the last vaccination intervals ≥ 14 days and the last attenuated live vaccine intervals≥28days
6. temperature ≤ 37℃

Inclusion criteria for group Ⅳ（JE-L+EV71）were as follows:

1. aged ≥ 8 months
2. sign the informed consent form
3. the legal guardians participate in all the planned follow-up and be able to comply with all research procedures
4. there is no inoculation history of EV71 vaccine, and there is no history of EV71 infection
5. the last vaccination intervals ≥ 14 days and the last attenuated live vaccine intervals ≥ 28 days
6. temperature ≤ 37℃

Exclusion Criteria:

Exclusion criteria for first needle:

1. the history or family history of anaphylaxis, convulsion, epilepsy, encephalopathy and psychosis
2. the history of severe inoculation allergies
3. patients with immunodeficiency and malignant tumors during the treatment period, receiving immunosuppressive therapy (oral steroid) or HIV due to low immunity, or family members have congenital immune disease
4. Nonspecific immunoglobulin was injected within one month
5. temperature≥37.1℃ and infectious diseases
6. the history of thrombocytopenia or other thrombocytopenia with a definite diagnosis
7. respiratory disease, acute infection or chronic disease activity period
8. severe cardiovascular disease, liver and kidney disease, and complications of diabetes
9. infectious, suppurative and allergic dermatosis
10. other conditions that may affect the evaluation of the trail

Exclusion criteria for follow-up needle:

1. any serious adverse events that have a causal relationship with the inoculation of the upper dose of the vaccine
2. the abnormality of 4 levels (local, systemic adverse reactions and vital signs) was judged to be related to vaccination
3. other new standards of exclusion criteria for first needle
4. other conditions that may affect the evaluation of the trail

Ages: 6 Months to 12 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1944 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2019-04 (Estimated)

PRIMARY OUTCOMES:
Antibody positive rate to vaccinations | within 90 days after the last vaccination
  The definition of EV71 vaccine positive for antibody titers <1:8 before inoculation, antibody titers ≥ 1:8 after inoculation; or before inoculation antibody titer is above 1:8,the titer after vaccination appeared more than 4 times growth.Hepatitis B vaccine seroconversion was defined as Anti-HBs<10mIU/ml before inoculation, Anti-HBs after inoculation was more than 10mIU/ml.Leprosy vaccine using ELISA detection test, measles >200U/ml positive for rubella >20U/ml positive or positive before inoculation, antibody positive growth is more than 4 times.Japanese encephalitis vaccine using PRNT test before immunization antibody titer after inoculation was less than 1:5, at 1:10, or after vaccination antibody titer than before inoculation is no less than 4 times of growth is positive. A meningococcal bactericidal antibody level in serum by micro bactericidal antibody test, the antibody titer after inoculation than before inoculation is more than 4 times growth is positive.
Antibody titer / concentration to vaccination | within 90 days after the last vaccination
  Blood samples from the participants were collected before and after vaccination, the changes of serum concentration and titer were determined by serum test.

SECONDARY OUTCOMES:
Number of Participants at the Injection Site, Solicited Systemic Reactions, or Any Unsolicited Adverse Events | within 90 days after the last vaccination
  Participants were provided with diary cards to record the occurrence and severity of solicited local reactions at the injection site (pain, induration, erythema, edema, pruritus) during 7 days after vaccination, solicited systemic reactions (fever, headache, fatigued, cough, myalgia, asthenia, vertigo, diarrhea), and any unsolicited adverse during 29 days after vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong Provincial Center for Disease Control and Prevention, Jinan, Shandong, China

REFERENCES:
- [Derived] Liu X, Chang S, Wang R, Xiao Y, Li F, Xu Q, Zhang S, Chen X, Zhang S, Zhang M, Chen X, Cao Q, Liu X, Wang H, Zhan D, Chen H, Chen W, Jiang J, Zhang C, Wang H, Gao L, Shi X, Yang X, Xu A. Immunogenicity and Safety of an Inactivated Enterovirus 71 Vaccine Administered Simultaneously with Hepatitis B Virus Vaccine, Group A Meningococcal Polysaccharide Vaccine, Measles-Rubella Combined Vaccine and Japanese Encephalitis Vaccine: A Multi-Center, Randomized, Controlled Clinical Trial in China. Vaccines (Basel). 2022 Jun 2;10(6):895. doi: 10.3390/vaccines10060895. PMID 35746502

DOCUMENTS (3):
  • Study Protocol (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT03519568/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-05): https://cdn.clinicaltrials.gov/large-docs/68/NCT03519568/SAP_001.pdf
  • Informed Consent Form (2017-10-27): https://cdn.clinicaltrials.gov/large-docs/68/NCT03519568/ICF_002.pdf